CLINICAL TRIAL: NCT04141332
Title: Specific Language Impairment (SLI) in Children May Caused by Epileptic Brain Activity
Status: Completed | Type: Observational
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Esmael, Assistant Prof of Neurology, Mansoura University Hospital
Other Study IDs: Mansoura University Hospital
Record Dates: First submitted 2019-10-23; First posted 2019-10-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Specific Language Impairment
MeSH Terms: conditions — Specific Language Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: 80 Patient
  Interventions: Diagnostic Test: EEG was recorded by EEG Machines
- Group 2: 80 Control subject
  Interventions: Diagnostic Test: EEG was recorded by EEG Machines

INTERVENTIONS:
Diagnostic Test: EEG was recorded by EEG Machines — EEG was recorded by EEG Machines

SUMMARY:
The objective of this study was to find if there is a possible association and the impact of epilepsy and epileptiform activity in children with SLI.

DETAILED DESCRIPTION:
This study concentrates on the impact of epileptiform activity for childhood epilepsy on the speech and language disturbances in addition to the associated social, cognitive and intellectual dysfunctions.

ELIGIBILITY:
Inclusion Criteria:

* 80 children were suffering from specific language impairment
* 80 healthy children with age and sex match control group.

Exclusion Criteria:

* Previous history of perinatal hypoxic-ischemic damage
* meningitis or encephalitis
* motor weakness
* hearing disorders
* IQ below seventy
* CP, social deprivation
* autism and
* psychiatric disorders .

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study was conducted on 80 children with speech disorders in preschool children.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
EEGs finding | 24-48 hours
  EEGs finding were defined according to the followings "Normal: within the range of frequency and amplitude distribution." "Epileptiform: Describes transient background activity with a characteristic spikes, sharp waves, spike-slow wave or sharp-slow wave complexes of focal or generalized distribution".
  "Abnormal non-epileptiform: deviations from normal in terms of background frequency patterns, usually in the form of excessive slow activity".

OTHER OUTCOMES:
Intelligence quotient (IQ) | 24-72 hours
  An intelligence quotient (IQ) is a total score derived from several standardized tests designed to assess human intelligence. Historically, IQ is a score obtained by dividing a person's mental age score, obtained by administering an intelligence test, by the person's chronological age, both expressed in terms of years and months. The resulting fraction is multiplied by 100 to obtain the IQ score.
  When current IQ tests were developed, the median raw score of the norming sample is defined as IQ 100 and scores each standard deviation (SD) up or down are defined as 15 IQ points greater or less.
social age | 24-48 hours
  Evaluation of social age: using the Vineland Social Maturity Scale . VSMS was used along with a cognitive assessment to help make a diagnosis of mental retardation or intellectual disability. It has also been used extensively to assess the development of activities of everyday life.
cognitive age | 24-48 hours
  Evaluation of cognitive age (mental age): using the Stanford Binet Intelligence Scale. The Stanford-Binet test is a examination meant to gauge intelligence through five factors of cognitive ability. These five factors include fluid reasoning, knowledge, quantitative reasoning, visual-spatial processing and working memory. Both verbal and nonverbal responses are measured.
language assessment | 24-72 hours
  Language evaluation: by Comprehensive Arabic Language Test (CALT). The CALT was constructed by the members of the Department of Phoniatrics at Alexandria Main University Hospital, Egypt, to form a detailed comprehensive assessment battery for Arabic language and test its reliability and validity to use it in the early detection of subtle changes in the various components of language in cases of language impaired children.

CONTACTS AND LOCATIONS:
Overall Officials: Esmael M Ahmed, MD, Principal Investigator — Assistant Prof of Neurology
Locations (1):
- Mansoura University Hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tomas E, Vissers C. Behind the Scenes of Developmental Language Disorder: Time to Call Neuropsychology Back on Stage. Front Hum Neurosci. 2019 Jan 9;12:517. doi: 10.3389/fnhum.2018.00517. eCollection 2018. PMID 30687040
- [Result] 2-Kraft, S.J. & De Thorne, L.S. The Brave New World of Epigenetics: Embracing Complexity in the Study of Speech and Language Disorders Current Developmental Disorders Reports . 2014; 1: 207.
- [Result] 3-Hillert, Dieter. Encyclopedia of Evolutionary Psychological Science, Chapter: Neurobiology of Language, Publisher: Springer, Editors Viviana Weekes-Shackelford, Todd K. Shackelford, Viviana A. Weekes-Shackelford. Neurobiology of Language.2016: pp.1-15
- [Result] Laasonen M, Smolander S, Lahti-Nuuttila P, Leminen M, Lajunen HR, Heinonen K, Pesonen AK, Bailey TM, Pothos EM, Kujala T, Leppanen PHT, Bartlett CW, Geneid A, Lauronen L, Service E, Kunnari S, Arkkila E. Understanding developmental language disorder - the Helsinki longitudinal SLI study (HelSLI): a study protocol. BMC Psychol. 2018 May 21;6(1):24. doi: 10.1186/s40359-018-0222-7. PMID 29784061
- [Result] Ghandour H, Eldin SK, Sallam Y, Mahmoud S. Associated comorbidities of specific language impairment. Benha Med J. 2018; 35:115-21.
- [Result] Carol Westby. Social-Emotional Outcomes for Children With SLI . Word of Mouth. 2017 ; 28 (4):1-5.
- [Result] Kim EH, Ko TS. Cognitive impairment in childhood onset epilepsy: up-to-date information about its causes. Korean J Pediatr. 2016 Apr;59(4):155-64. doi: 10.3345/kjp.2016.59.4.155. Epub 2016 Apr 30. PMID 27186225
- [Result] Syam UK, Thomas SV. Epileptiform activity in the electroencephalogram of 6-year-old children of women with epilepsy. Ann Indian Acad Neurol. 2016 Jul-Sep;19(3):318-22. doi: 10.4103/0972-2327.179974. PMID 27570381
- [Result] Holmes GL. What is more harmful, seizures or epileptic EEG abnormalities? Is there any clinical data? Epileptic Disord. 2014 Oct;16 Spec No 1(Spec No 1):S12-22. doi: 10.1684/epd.2014.0686. PMID 25323031
- [Result] Ung H, Cazares C, Nanivadekar A, Kini L, Wagenaar J, Becker D, Krieger A, Lucas T, Litt B, Davis KA. Interictal epileptiform activity outside the seizure onset zone impacts cognition. Brain. 2017 Aug 1;140(8):2157-2168. doi: 10.1093/brain/awx143. PMID 28666338
- [Result] McTague A, Howell KB, Cross JH, Kurian MA, Scheffer IE. The genetic landscape of the epileptic encephalopathies of infancy and childhood. Lancet Neurol. 2016 Mar;15(3):304-16. doi: 10.1016/S1474-4422(15)00250-1. Epub 2015 Nov 17. PMID 26597089
- [Result] Staley K. Molecular mechanisms of epilepsy. Nat Neurosci. 2015 Mar;18(3):367-72. doi: 10.1038/nn.3947. Epub 2015 Feb 24. PMID 25710839
- [Result] Faught E, Karakis I, Drane DL. The Impact of Interictal Discharges on Performance. Curr Neurol Neurosci Rep. 2018 Oct 8;18(12):88. doi: 10.1007/s11910-018-0892-9. PMID 30298240
- [Result] Luz-Escamilla L, Morales-Gonzalez JA. Association between Interictal Epileptiform Discharges and Autistic Spectrum Disorder. Brain Sci. 2019 Jul 30;9(8):185. doi: 10.3390/brainsci9080185. PMID 31366163
- [Result] Kane N, Acharya J, Benickzy S, Caboclo L, Finnigan S, Kaplan PW, Shibasaki H, Pressler R, van Putten MJAM. A revised glossary of terms most commonly used by clinical electroencephalographers and updated proposal for the report format of the EEG findings. Revision 2017. Clin Neurophysiol Pract. 2017 Aug 4;2:170-185. doi: 10.1016/j.cnp.2017.07.002. eCollection 2017. No abstract available. Erratum In: Clin Neurophysiol Pract. 2019 Jun 15;4:133. doi: 10.1016/j.cnp.2019.06.001. PMID 30214992
- [Result] Ghacibeh GA, Fields C. Interictal epileptiform activity and autism. Epilepsy Behav. 2015 Jun;47:158-62. doi: 10.1016/j.yebeh.2015.02.025. Epub 2015 Apr 3. PMID 25847431
- [Result] Shweta Singh, Shivani Pandey, Vivek Agarwal. A Comparative study of Vineland Adaptive Behavior Scale II and Vineland Social Maturity Scale on children and adolescents with Intellectual Disability J. Indian Assoc. Child Adolesc. Ment. Health 2019; 15(1):27-38.
- [Result] El-Maghraby R. Comprehensive Arabic Language test as a tool for assessing delayed language impaired Egyptian children [MD thesis]. Alexandria: Faculty of Medicine, Alexandria University;2008.
- [Result] Moreno MA. Speech and Language Delays in Young Children. JAMA Pediatr. 2015 Aug;169(8):796. doi: 10.1001/jamapediatrics.2014.2146. No abstract available. PMID 26237464
- [Result] Fadhli, Khadija & Al-Bunaian, Nada. Prevalence and Social Influences of Delayed Language Development in Preschool-Age Saudi Children. International Journal of Science and Research. 2017:6. 6-391.
- [Result] Wallace IF, Berkman ND, Watson LR, Coyne-Beasley T, Wood CT, Cullen K, Lohr KN. Screening for Speech and Language Delay in Children 5 Years Old and Younger: A Systematic Review. Pediatrics. 2015 Aug;136(2):e448-62. doi: 10.1542/peds.2014-3889. Epub 2015 Jul 7. PMID 26152671
- [Result] Reilly S, Tomblin B, Law J, McKean C, Mensah FK, Morgan A, Goldfeld S, Nicholson JM, Wake M. Specific language impairment: a convenient label for whom? Int J Lang Commun Disord. 2014 Jul-Aug;49(4):416-51. doi: 10.1111/1460-6984.12102. PMID 25142091
- [Result] Kalnak N, Peyrard-Janvid M, Sahlen B, Forssberg H. Family history interview of a broad phenotype in specific language impairment and matched controls. Genes Brain Behav. 2012 Nov;11(8):921-7. doi: 10.1111/j.1601-183X.2012.00841.x. Epub 2012 Sep 20. PMID 22928858
- [Result] Baumer FM, Cardon AL, Porter BE. Language Dysfunction in Pediatric Epilepsy. J Pediatr. 2018 Mar;194:13-21. doi: 10.1016/j.jpeds.2017.10.031. Epub 2017 Dec 11. No abstract available. PMID 29241678
- [Result] Tuchman R. Autism and Cognition Within Epilepsy: Social Matters. Epilepsy Curr. 2015 Jul-Aug;15(4):202-5. doi: 10.5698/1535-7511-15.4.202. PMID 26316868
- [Result] Hamdy M. Bedair, Mona K. Mohamed, Rania M. Abdou, Faten I. El Kafrawy. Concurrent language disorders in children with idiopathic epilepsy. Egyptian Journal of Otolaryngology. 2017: 33 (3): 603-609.
- [Result] Mehta B, Chawla VK, Parakh M, Parakh P, Bhandari B, Gurjar AS. EEG Abnormalities in Children with Speech and Language Impairment. J Clin Diagn Res. 2015 Jul;9(7):CC04-7. doi: 10.7860/JCDR/2015/13920.6168. Epub 2015 Jul 1. PMID 26417549
- [Result] Jones JE, Siddarth P, Gurbani S, Shields WD, Caplan R. Cognition, academic achievement, language, and psychopathology in pediatric chronic epilepsy: Short-term outcomes. Epilepsy Behav. 2010 Jul;18(3):211-7. doi: 10.1016/j.yebeh.2010.03.015. Epub 2010 May 14. PMID 20471326
- [Result] Sanchez Fernandez I, Loddenkemper T, Galanopoulou AS, Moshe SL. Should epileptiform discharges be treated? Epilepsia. 2015 Oct;56(10):1492-504. doi: 10.1111/epi.13108. Epub 2015 Aug 21. PMID 26293670
- [Result] Parry-Fielder B, Collins K, Fisher J, Keir E, Anderson V, Jacobs R, Scheffer IE, Nolan T. Electroencephalographic abnormalities during sleep in children with developmental speech-language disorders: a case-control study. Dev Med Child Neurol. 2009 Mar;51(3):228-34. doi: 10.1111/j.1469-8749.2008.03163.x. Epub 2009 Jan 29. PMID 19207301